CLINICAL TRIAL: NCT05075278
Title: Assessing the Quality and Effectiveness of Two Common Supervision Models in Training Environments Using a Validated Supervision Instrument
Brief Title: Supervision Models in Training Environments
Acronym: VSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1734757
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Supervision; Anesthesia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attending physician for direct 1:1 supervision (Active Comparator): Participants will be assigned to an attending physician for direct 1:1 supervision. The participants will fill out a survey at the end of the day for 16 consecutive days.
  Interventions: Behavioral: Survey
- Senior resident for direct 1:1 supervision (Experimental): Participants will be assigned to an senior resident as a direct supervisor with oversight from an attending physician (in accordance with CMS/ACGME staffing criteria). The participants will fill out a survey at the end of the day for 16 consecutive days.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — A survey will be completed by the participants at the conclusion of each day.

SUMMARY:
Attending physicians often supervise novice junior residents in a direct one-to-one format. Alternatively, a senior resident can be paired with a new trainee under the non-direct (but immediately available) supervision of an attending physician. Resident supervision has been considered an important step towards independent practice. Both models are ubiquitous in the United States, but no study to date has been performed if one model is better than the other with respect to supervision scores.

DETAILED DESCRIPTION:
Supervision of residents is a cornerstone of ACGME accreditation and a critical focus of any training program. A nine-faceted, validated survey has been used to assess quality and effectiveness of supervision in training environments. Residents that assign poor scores for faculty members also tend to poorly evaluate the department-at-large. Further, residents that evaluate supervisors unfavorably also tend to report more patient safety mishaps in the context of a less safe work environment. Previous literature that used this supervision scale concluded that residents who reported mean department-wide supervision scores less than 3 (frequent) reported significantly more frequent occurrences of mistakes with negative consequences to patients and medication errors.

Attending physicians often supervise novice junior residents in a direct one-to-one format. Alternatively, a senior resident can be paired with a new trainee under the non-direct (but immediately available) supervision of an attending physician. Resident supervision has been considered an important step towards independent practice.. Both models are ubiquitous in the United States, but no study to date has been performed if one model is better than the other with respect to supervision scores.

ELIGIBILITY:
Inclusion Criteria:

* New incoming anesthesia residents assigned to healthy patients (ASA physical status classifications of 1 or 2).

Exclusion Criteria:

* New incoming anesthesia residents assigned to patients with ASA physical status classifications 3 or greater.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Supervision evaluation questionnaire | At the conclusion of each day for 16 consecutive days
  A series of questions pertaining to planning perianesthesia care, feedback, availability, opportunities, stimulating patient based learning, professionalism, interpersonal skills, presence, and safety. It questions are scored using a 4-point Likert scale (never = 1, rarely = 2, frequently = 3, and always = 4). A score less than 3 is associated with more frequent occurrences of mistakes.

SECONDARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory Short Form | At the conclusion of each day for 16 consecutive days
  (Strongly agree=5, Agree=4, Neither=3, Disagree=2, Strongly Disagree=1).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Malgieri, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Oliveira GS Jr, Rahmani R, Fitzgerald PC, Chang R, McCarthy RJ. The association between frequency of self-reported medical errors and anesthesia trainee supervision: a survey of United States anesthesiology residents-in-training. Anesth Analg. 2013 Apr;116(4):892-7. doi: 10.1213/ANE.0b013e318277dd65. Epub 2013 Feb 5. PMID 23385057
- [Background] De Oliveira GS Jr, Dexter F, Bialek JM, McCarthy RJ. Reliability and validity of assessing subspecialty level of faculty anesthesiologists' supervision of anesthesiology residents. Anesth Analg. 2015 Jan;120(1):209-213. doi: 10.1213/ANE.0000000000000453. PMID 25268396
- [Background] Riveros Perez E, Jimenez E, Yang N, Rocuts A. Evaluation of Anesthesiology Residents' Supervision Skills: A Tool to Assess Transition Towards Independent Practice. Cureus. 2019 Feb 26;11(2):e4137. doi: 10.7759/cureus.4137. PMID 31058020
- [Result] de Oliveira Filho GR, Dal Mago AJ, Garcia JH, Goldschmidt R. An instrument designed for faculty supervision evaluation by anesthesia residents and its psychometric properties. Anesth Analg. 2008 Oct;107(4):1316-22. doi: 10.1213/ane.0b013e318182fbdd. PMID 18806047